CLINICAL TRIAL: NCT03936543
Title: Comparison of the Needle Tip Location According to the Position of the Operator During Short Axis Ultrasound Guided Central Venous Catheterization in the Left Internal Jugular Vein
Brief Title: Comparison of the Needle Tip Location by the Position of the Operator During Ultrasound Guided LIJV Catheterization.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Kyong Kim, Clinical assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 20190311/10-2019-7/041
Record Dates: First submitted 2019-05-02; First posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Catheterization, Central Venous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended axillary midline (Experimental): Operator stands at the bedside on extended midline of the patient's lt. axilla during lt. internal jugular vein catheterization
  Interventions: Other: Position change
- Extended head midline (Active Comparator): Operator stands at the bedside on extended midline of the patient's head during lt. internal jugular vein catheterization.
  Interventions: Other: Conventional position

INTERVENTIONS:
Other: Position change — Different position during central line catheterization
  Arms: Extended axillary midline
Other: Conventional position — Conventional position during central line catheterization
  Arms: Extended head midline

SUMMARY:
When the left internal jugular vein catheterization under short-axis ultrasound guided, an operator should be stand around the lying patient's head. The investigators are going to evaluate to effects of the operator's location.

DETAILED DESCRIPTION:
When placing the central line catheter in the left internal jugular vein under short-axis ultrasound guided, an operator should be stand around the lying patient's head. The investigators are going to evaluate to effects of the operator's location. (Above the midline of patient's head versus above the left extended axillary line)

ELIGIBILITY:
Inclusion Criteria:

* Central venous catheterization required on lt. IJV

Exclusion Criteria:

* History of cervical spine surgery
* Abnormal structure of cervical spine, carotid artery or jugular vein
* Disease of carotid artery
* Immobilization due to cervical spine fracture or other diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Distance from needle tip to center of IJV | intraoperative
  The distance that the needle tip is placed from the center of the jugular vein when the needle is fixed after the vascular puncture

CONTACTS AND LOCATIONS:
Overall Officials: Tae Kyong Kim, MD, phD, Study Director — SMG-SNU Boramae hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ishizuka M, Nagata H, Takagi K, Kubota K. Right internal jugular vein is recommended for central venous catheterization. J Invest Surg. 2010 Apr;23(2):110-4. doi: 10.3109/08941930903469342. PMID 20497014
- [Background] Lobato EB, Sulek CA, Moody RL, Morey TE. Cross-sectional area of the right and left internal jugular veins. J Cardiothorac Vasc Anesth. 1999 Apr;13(2):136-8. doi: 10.1016/s1053-0770(99)90075-7. PMID 10230944
- [Background] Sulek CA, Blas ML, Lobato EB. A randomized study of left versus right internal jugular vein cannulation in adults. J Clin Anesth. 2000 Mar;12(2):142-5. doi: 10.1016/s0952-8180(00)00129-x. PMID 10818329
- [Background] Lieberman JA, Williams KA, Rosenberg AL. Optimal head rotation for internal jugular vein cannulation when relying on external landmarks. Anesth Analg. 2004 Oct;99(4):982-988. doi: 10.1213/01.ANE.0000132908.77111.CA. PMID 15385337
- [Derived] Min SW, Kim H, Won D, Chang JE, Lee JM, Hwang JY, Kim TK. Comparison of the needle tip location with the operator's position during ultrasound-guided internal jugular vein catheterization: A randomized controlled study. Medicine (Baltimore). 2022 Oct 28;101(43):e31249. doi: 10.1097/MD.0000000000031249. PMID 36316874